CLINICAL TRIAL: NCT06507969
Title: The Effect of Body Composition on Respiratory Parameters, Functional Capacity and Sleep in Healthy Young Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Kent University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melis Usul, Research Assistant, Istanbul Kent University
Other Study IDs: IstanbulKentU-FTR-MU-02
Record Dates: First submitted 2024-07-07; First posted 2024-07-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Body Weight
Keywords: body composition; Respiratory Function Tests; Sleep Quality
MeSH Terms: conditions — Body Weight; Sleep Initiation and Maintenance Disorders | interventions — Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young adults aged 18-30 years: Sociodemographic information of all participants will be obtained within the scope of the evaluations. Body composition parameters will be measured with Tanita DC360 Body Analysis Scale. In pulmonary function test, Forced vital capacity (FVC), Forced expiratory volume in 1st second (FEV1), Tiffeneau ratio (FEV1/FVC), peak expiratory flow rate (PEF) values will be evaluated with COSMED Pony FX (COSMED; Italy) spirometer. Respiratory muscle endurance will be assessed by Maximum Minute Ventilation will be determined. Pittsburg Sleep Quality, a reliable questionnaire that assesses sleep quality The index will be filled in by the participants. 6 Minutes to assess functional capacity A walking test will be performed and the distance travelled by individuals will be recorded.
  Interventions: Other: The Effect of Body Composition on Respiratory Parameters, Functional Capacity and Sleep in Healthy Young Adults

INTERVENTIONS:
Other: The Effect of Body Composition on Respiratory Parameters, Functional Capacity and Sleep in Healthy Young Adults — Sociodemographic information of all participants will be obtained within the scope of the evaluations. Body composition parameters will be measured with Tanita DC360 Body Analysis Scale. In pulmonary function test, Forced vital capacity (FVC), Forced expiratory volume in 1st second (FEV1), Tiffeneau ratio (FEV1/FVC), peak expiratory flow rate (PEF) values will be evaluated with COSMED Pony FX (COSMED; Italy) spirometer. Respiratory muscle endurance will be assessed by Maximum Minute Ventilation will be determined. Pittsburg Sleep Quality, a reliable questionnaire that assesses sleep quality The index will be filled in by the participants. 6 Minutes to assess functional capacity A walking test will be performed and the distance travelled by individuals will be recorded

SUMMARY:
Body composition has a significant effect on the respiratory system. Both respiratory prediction of function and a prognostic tool evaluated in the cardiopulmonary system factor. Respiratory function, which directly affects respiratory muscle strength and respiratory muscle endurance covers a range of data. In the literature, the relationship between body composition and respiratory function. Although there are studies examining body composition in healthy young adults, the relationship between them has not been clearly demonstrated.

The aim of the study was to investigate the effects of body composition on respiratory function, respiratory muscle endurance, functional capacity and sleep quality.

For this purpose, at least 46 healthy young participants who fulfil the inclusion criteria will participate in the evaluation. Body composition parameters will be measured by the researchers using Tanita DC360 Body Analysis Scale. In pulmonary function test, forced vital capacity (FVC), forced expiratory volume in 1st second (FEV1), Tiffeneau ratio (FEV1/FVC), peak expiratory flow rate (PEF) values will be evaluated by the researchers with COSMED Pony FX (COSMED; Italy) spirometer and respiratory muscle endurance with Maximum Voluntary Ventilation test. Participants will answer the Pittsburg Sleep Quality Index. The 6-minute walk test will be applied to the participants with the instructions of the researchers.

Data will be analysed by SPSS Statistical Package for Social Sciences (SPSS) Version 20.0 (SPSS Inc., Chicago, Illinois) programme will be made using.

DETAILED DESCRIPTION:
Body composition is an important determinant of health and can be used in the assessment of cardiopulmonary problems. Body mass index (BMI) in cardiopulmonary function is an independent prognostic factor. Fat and lean mass have also been identified as strong predictors of physical fitness and mortality.

Pulmonary function is a long-term determinant of all-cause mortality, particularly cardiovascular mortality. Pulmonary function may be affected by malnutrition, recurrent.

It may be influenced by various genetic or environmental factors such as infections and exposure to toxic substances, obesity and systemic diseases.Pulmonary function testing is one of the basic and essential tests for the diagnosis and evaluation of lung diseases such as lung dysfunction, chronic obstructive pulmonary disease (COPD) and asthma. Factors affecting pulmonary function include age, body weight and height, and gender. Since these factors are significantly related to pulmonary function, they are used to calculate the regression equation and predicted normal values of the pulmonary function test.

The correlation between body mass index (BMI), waist size, fat mass and pulmonary function has been studied since the late 1950s. However, the correlation between pulmonary function and body The study results of the correlation between body composition and respiratory function were found to be different from each other. In addition, the mechanism by which body composition affects respiratory function is not fully understood.

Obesity and thus abdominal adiposity also affect aerobic capacity, respiratory function and respiratory muscle strength. Fat accumulation on the chest and abdominal walls inhibits the movement of the respiratory muscles, increases pleural pressure and reduces lung compliance, resulting in a decrease in the compliance of the respiratory system as a whole. Due to all these causes, decreases in functional residual capacity, expiratory reserve volume, forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and respiratory muscle strength are observed.

Strength and endurance tests are recommended to determine decreases in respiratory muscle performance.

Although the number of studies examining the relationship between respiratory muscle strength and body composition is higher in the literature, it has been shown that endurance assessment is more functionally meaningful because inspiratory muscles are used at submaximal level in daily life activities.

Sleep quality is associated with many factors such as age, gender, genetic and environmental factors, social life, economic status, stress, pain, substance abuse, physical diseases, physical activity level, eating habits and obesity.

In the literature, there are many studies examining the relationship between obesity and sleep quality using body composition parameters such as Body Mass Index (BMI), waist circumference, waist-to-hip ratio, and body fat percentage. In some of these studies, it has been suggested that there is no relationship between obesity and sleep quality; in others, it has been shown that obesity is associated with sleep problems, this relationship can be explained by a bidirectional mechanism, sleep problems such as poor sleep quality lead to obesity due to abnormal changes in metabolic and endocrine functions, and obesity leads to various pathological conditions associated with respiration. Obstructive sleep apnoea and obesity hypoventilation syndrome are among these conditions. Therefore, body composition has a significant effect on sleep quality and thus respiratory parameters.

In the literature, there are studies examining the relationship between body composition and respiratory function and respiratory muscle strength in healthy young adults. However, there is no study in the literature investigating the relationship between body composition and respiratory muscle endurance, functional capacity, respiratory function and sleep quality. The aim of study was to investigate the effect of body composition on respiratory function, respiratory muscle strength, respiratory muscle endurance and functional capacity in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer young adults between the ages of 18-30 who are willing to participate in the study
* Providing independent ambulation
* Individuals without cognitive/mental problems

Exclusion Criteria:

* Lack of co-operation
* Presence of diseases affecting the cardiac and pulmonary system
* Those with a history of neurological, rheumatic or metabolic diseases
* Pregnant women
* Presence of major musculoskeletal problems
* Individuals who smoke

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteer young adults between the ages of 18-30 who are willing to participate in the study
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Body composition | 10 minute
  The body analyses of the participants were performed by the bioelectrical impedance analysis technique by the researchers using "Tanita DC 360 Body Analyser Scale". Body mass index (kg/m2), muscle mass (kg), bone mass (kg) will be recorded by the researchers.
Respiratory parameters | 10 minute
  Pulmonary function test is a test used to evaluate respiratory parameters.Pulmonary function test was planned by COSMED Pony FX in accordance with the American Thoracic Society and European Respiratory Society criteria. Forced vital capacity, forced expiratory volume in 1st second , Tiffeneau ratio (FEV1/FVC), peak expiratory flow rate values and percentage of predictive values will be recorded by the investigators.
  Maximum Voluntary Ventilation test will be applied by the researchers to determine the respiratory muscle endurance of the participants.

SECONDARY OUTCOMES:
Functional Capacity | 6 minute
  The 6-minute walk test is a test that determines functional capacity. Participants will walk along a 30 metre straight corridor for 6 minutes.The distance covered by walking as fast as possible without running will be recorded by the investigators in metres.
Pittsburg Sleep Quality Indeks | 5 minute
  Pittsburg Sleep Quality Index developed is a questionnaire that evaluates sleep quality. It will be used to evaluate the sleep quality of the participants. The scale consists of 24 questions in total. Sleep duration, subjective sleep quality, time to fall asleep, effectiveness of habitual sleep, presence of sleep disorders, use of medication to fall asleep and daytime sleep dysfunction.
  Each item of the scale is evaluated between 0-3 points; the sum of the scores of the seven subcomponents gives the total score of the scale. The lowest score that can be obtained from the scale is 0 and the highest score is 21. A total score greater than 5 indicates that the sleep quality of the individual is not good.

CONTACTS AND LOCATIONS:
Overall Officials: Melis USUL, RA., Principal Investigator — Istanbul Kent University
Locations (1):
- Istanbul Kent University, Istanbul, Kagıthane-Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No